CLINICAL TRIAL: NCT06246136
Title: A Prospective, Multicenter, Randomized Clinical Trial to Evaluate the Safety and Effectiveness of ELIOS vs Competitor in Patients With Open-Angle Glaucoma Undergoing Cataract Surgery
Brief Title: Comparative Effectiveness and Safety of ELIOS in Patients With Open-Angle Glaucoma Undergoing Cataract Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elios Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELIOS-RCT STERLING
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Open Angle Glaucoma
Keywords: Excimer Laser; Micro-bypass; Trabeculostomy
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): ELIOS
  Interventions: Procedure: ELIOS
- Arm 2 (Active Comparator): Competitor Device
  Interventions: Procedure: Competitor Device

INTERVENTIONS:
Procedure: ELIOS — Following cataract surgery, surgeon will proceed to ELIOS treatment.
  Arms: Arm 1
Procedure: Competitor Device — Following cataract surgery, surgeon will proceed to Competitor treatment.
  Arms: Arm 2

SUMMARY:
The primary study objective is to compare the effectiveness of the combination of phacoemulsification with intraocular lens implant with ELIOS or competitor device in reducing IOP at 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects.
2. 40 years old or older.
3. Diagnosis of mild to moderate primary open-angle glaucoma, pseudoexfoliation glaucoma or pigmentary glaucoma:
4. Visually significant cataract eligible for phacoemulsification.

Exclusion Criteria:

1. All forms of angle closure glaucoma
2. Secondary glaucoma, including traumatic, neovascular, uveitic, lens-induced, steroid-induced, angle-recession, glaucoma associated with vascular disorders, and glaucoma associated with increased episcleral venous pressure
3. Congenital or developmental glaucoma
4. Prior incisional glaucoma surgery, intraocular surgery or ocular laser treatment of any type with the exception of selective laser trabeculoplasty (SLT) occurring a minimum of 6 months prior to the Screening visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
PRIMARY EFFECTIVENESS ENDPOINTS : IOP | 12 months
  Mean change in post-washout diurnal IOP from baseline to 12 months.

SECONDARY OUTCOMES:
SECONDARY EFFECTIVENESS ENDPOINTS : Post-washout diurnal IOP | 24 months
  Proportion of patients achieving 20% reduction in post-washout diurnal IOP from baseline.
SECONDARY EFFECTIVENESS ENDPOINTS : Number of hypotensive medications | 12 months
  change in number of hypotensive medications from screening to 12 months
SECONDARY EFFECTIVENESS ENDPOINTS : Treated IOP | 12 months
  Mean change in treated IOP from screening to 12 months
SECONDARY EFFECTIVENESS ENDPOINTS : Medications | 12 months
  Proportion of patients Medication free at 12 months

OTHER OUTCOMES:
SAFETY ENDPOINTS : adverse events | 24 months
  Rates of ocular adverse events
Safety endpoints: Retinal nerve fiber layer thickness | 12 months (with a planned extension of analysis at 24 months)
  measurement of Retinal nerve fiber layer thickness

CONTACTS AND LOCATIONS:
Locations (16):
- ELIOS Clinical Site, Leuven, Belgium
- France (3):
  - Elios Clinical Site, Avranches
  - ELIOS Clinical Site, Bordeaux
  - ELIOS clinical site, Paris
- Germany (3):
  - ELIOS Clinical Site, Bochum
  - Elios clinical site, Bonn
  - ELIOS clinical site, Heidelberg
- ELIOS Clinical Site, Maastricht, Netherlands
- Spain (3):
  - ELIOS clinical site, Barcelona
  - ELIOS Clincal Site, Madrid
  - ELIOS Clinical site, Madrid
- United Kingdom (5):
  - ELIOS Clinical Site, East Grinstead
  - ELIOS Clinical Site, Edinburgh
  - ELIOS Clinical Site, Guildford
  - ELIOS clinical site, London
  - ELIOS Clinical Site, Manchester

IPD SHARING:
Plan to Share IPD: Undecided